CLINICAL TRIAL: NCT03621579
Title: Analysis of Retinal Nerve Fiber Layer and Macular Thickness After Congenital Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, director, Wenzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNFL-HZ
Record Dates: First submitted 2018-04-10; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Congenital Cataract
Keywords: RNFLT
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the RNFLT and CMT (Other): the retinal nerve fiber layer (RNFLT) and macular thickness (CMT)
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — To measure the RNFLT and CMT in congenital cataracts before and after the cataract extraction with IOL implantation surgery

SUMMARY:
Congenital cataract is the main cause of form deprivation amblyopia in children. Current studies confirm that form deprivation amblyopia affects the retinal nerve fiber layer. However, there are different opinions about the effect of amblyopia on the optic nerve fiber thickness around the optic disc at home and abroad. Investigators have performed "cataract extraction with IOL implantation" on children with bilateral and unilateral congenital cataract. Investigators used OCT biometry to measure children's the retinal nerve fiber layer (RNFLT) and macular thickness (CMT) before and after surgery. Investigators dynamically observed changes in RNFL and CMT to explore the retinal mechanism of form deprivation amblyopia and help guide the clinical correct understanding of postoperative follow-up time.

DETAILED DESCRIPTION:
This prospective study reviewed children with CC who were undergoing cataract extraction with IOL implantation at the Eye Hospital of Wenzhou Medical University, Hangzhou, China. bilateral and unilateral CC children were placed in Study group, while age-matched normal children were included as controls. Children who were uncooperative to complete the preoperative and postoperative examinations were excluded.

All eyes were divided into 4 groups. Group 1: form deprivation amblyopia of unilateral CC, Group 2: unaffected eyes of unilateral CC, Group 3: form deprivation amblyopia of bilateral CC, Group 4: normal eyes of normal children. The preoperative and postoperative data including sex, age at surgery, 7 position of RNFLT and CMT were collected.

All surgeries were performed by the same surgeon (Y.E.Z.) under general anesthesia. Investigators used OCT biometry to measure participants' the retinal nerve fiber layer (RNFLT) and macular thickness (CMT) before surgery and 1 week, 1 month, 3 months, and 6 months and 1 year after surgery, and compared with age-matched normal children.

ELIGIBILITY:
Inclusion Criteria:

* congenital cataract

Exclusion Criteria:

* incooperative to complete the preoperative and postoperative examinations

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
RNFLT | 1 year
  the retinal nerve fiber layer thickness (RNFLT)measured by OCT biometry (Units :um)
CMT | 1 year
  the macular thickness (CMT) measured by OCT biometry (Units :um)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang
  - Ophthalmology and Optometry Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bansal P, Ram J, Sukhija J, Singh R, Gupta A. Retinal Nerve Fiber Layer and Macular Thickness Measurements in Children After Cataract Surgery Compared With Age-Matched Controls. Am J Ophthalmol. 2016 Jun;166:126-132. doi: 10.1016/j.ajo.2016.03.041. Epub 2016 Apr 5. PMID 27059633